CLINICAL TRIAL: NCT03647553
Title: The Nash-wo-Numa (Childhood Growth & Development) Study : Factors That Impact Linear Growth and Mental Health in Children 9-15 Years of Age in Matiari, Pakistan
Brief Title: The Nash-wo-Numa (Childhood Growth & Development) Study
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Collaborators: The Hospital for Sick Children (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Founding Director of the Center of Excellence in Women and Child Health, Aga Khan University
Other Study IDs: 5251-WCH-ERC-18
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Adolescent Development; Stunting; Depression; Micronutrient Deficiency
MeSH Terms: conditions — Growth Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — As described in the protocol. Blood specimen will be stored for future analysis of few assays, based on funding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The proposed study will be a cross-sectional study in the District of Matiari, Pakistan. Children ages 9-15 years will be identified from a Matiari District household census scheduled being conducted from December 2016- to May 2017 by the Department of Pediatrics and Child Health, Aga Khan University. Anthropometric measures, Tanner Stage, Hemoglobin concentration, blood draw as well as questionnaires will be assessed in all participants.

ELIGIBILITY:
Inclusion Criteria:

* All girls between 9.0-14.9 years of age and boys between 10.0-15.9 years of age at the time of enrollment who are permanent residents of Matiari are eligible to participate in the Nash-wo-Numa Study.
* The participant's birth mother must also be available to participate in the study and be cognitively able to answer questions since they will be able to provide more accurate information about the birth characteristics of the participant as well as household information like dietary intake

Exclusion Criteria:

* Children not meeting the age criteria will not be invited to participate in the study. Female participants who are pregnant or have been pregnant will be excluded from the study.
* Participants must not be participating in any other nutrition trials. Participants with known chronic or genetic diseases that impact growth will be excluded.
* An illustrative list of conditions include: congenital heart disease, metabolic disorders (e.g. diabetes), cancer, genetic disorders (Down's syndrome, Turner's syndrome), blood disorders (symptomatic thalassemia, sickle cell anaemia), chronic disorders (kidney i.e. nephrotic syndrome, gastrointestinal i.e. Crohn's, bone dysplasia, immunodeficiency disorders).

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted in Matiari District in the Province of Sindh, Pakistan. The population of Matiari (2017) was estimated to be 769,349 with approximately 85% being rural. There are approximately 48,000 school-aged children between 9.0 and 15.9 years of age living in the District, which is representative of rural conditions in Pakistan.
Sampling Method: Probability Sample
Enrollment: 1385 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Stunting | through study completion, an average of 1 year
  < -2 Height-for-age z-score

SECONDARY OUTCOMES:
Factors associated with impaired linear growth | through study completion, an average of 1 year
  To identify factors associated with impaired linear growth among girls between 9-14.9 years of age and boys 10-15.9 years of age living in Matiari
Anemia and micronutrient deficiencies | through study completion, an average of 1 year
  To determine the prevalence of anemia and micronutrient deficiencies among girls between 9-14.9 years of age and boys 10-15.9 years of age living in Matiari
Household Dietary Diversity Scale (HDDS) | through study completion, an average of 1 year
  The HDDS reflects household access to food variation and is a count of the food groups consumed over a given reference period. The value of this variable will range from 0 to 12 and represents the total number of food groups consumed.
Food Insecurity Experience Scale (FIES) | through study completion, an average of 1 year
  FIES was developed in 2013 by the FAO for global and country monitoring of the severity of food insecurity in the previous 12 months. Since 2014, the Gallup World Poll (GWP) has collected data using the FIES. The FIES consists of eight dichotomous questions and results range on a scale from mild to severe food insecurity. Results are classified based on the total number of affirmative responses ranging from 0-8. While the FIES does not measure food insecurity directly in children, estimates of the percentage of children living in food-insecure households are generally used.
Anxiety | through study completion, an average of 1 year
  To access the presalence of anxiety we will be using the Screen for Child Anxiety Related Disorders (SCARED). This instrument contains 41 items and measures anxiety using four domains: panic/somatic, separation anxiety, generalized anxiety, and school phobia. A total score >25 indicates an anxiety disorder.
Depression | through study completion, an average of 1 year
  To determine the prevalence of depression among girls between 9-14.9 years of age and boys 10-15.9 years of age living in Matiari. We will be using the Mood and Feeling questionnaire to assess depression. A score > 27 may indicate the presence of depression.
Pubertal status | through study completion, an average of 1 year
  To determine the prevalence of pubertal status (pre-puberty, in-puberty, completing puberty) according to chronological age among girls between 9-14.9 years of age and boys 10-15.9 years of age living in Matiari using culturally sensitive methods. Puberty assessment for this study will be composed of two components:
  1. Self-Assessment: All participants will be asked a series of questions similar to a medical history to determine their Pubertal Phase ;
  2. Physical Assessment: Participants also willing to participate in a modified physical examination for Tanner Stage assessment. Puberty Phase classification after Tanner Stage assessment. Study staff will confirm assent and consent for each physical Tanner Stage assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Matiari Research and Training Centre, Matiari, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Campisi SC, Humayun KN, Wasan Y, Soofi SB, Islam M, Hussain A, Shakeel A, Vandermorris A, Soder O, Bhutta ZA. The relationship between pubertal timing and under-nutrition in rural Pakistan. J Adolesc. 2021 Apr;88:58-66. doi: 10.1016/j.adolescence.2021.02.002. Epub 2021 Feb 19. PMID 33618265
- [Derived] Campisi SC, Wasan Y, Soofi S, Monga S, Korczak DJ, Lou W, Soder O, Vandermorris A, Humayun KN, Mian A, Szatmari P, Bhutta ZA. Nash-wo-Numa (childhood growth & development) study protocol: factors that impact linear growth in children 9 to 15 years of age in Matiari, Pakistan. BMJ Open. 2019 Jun 12;9(6):e028343. doi: 10.1136/bmjopen-2018-028343. PMID 31196903